CLINICAL TRIAL: NCT04627896
Title: Safety and Efficacy of a Novel 3D Cartography-based Targeted Microwave Focal Therapy Device in Men With Localized Low to Intermediate-risk Prostate Cancer
Brief Title: Targeted Microwave Focal Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Koelis (Industry)
Responsible Party: Principal Investigator, Marco Oderda, Principal Investigator, A.O.U. Città della Salute e della Scienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0005732
Record Dates: First submitted 2020-02-16; First posted 2020-11-13 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer Stage I
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Targeted microwave ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Katty focal therapy (Experimental): Patients fulfilling inclusion criteria undergo focal treatment with Trinity-guided Katty device
  Interventions: Device: Katty focal therapy

INTERVENTIONS:
Device: Katty focal therapy — Microwave ablation with TATO3 generator (Katty system) under guidance of ultrasound/mpMRI fusion image device Trinity

SUMMARY:
Focal therapy (FT) for prostate cancer (PCa) is an interesting therapeutic option for localized disease with a favorable low- to intermediate-risk profile. The aim of this approach is to offer a personalized and less aggressive treatment as compared to radical treatments such as radical prostatectomy (RP) or primary radiation therapy, reducing functional morbidity while maintaining oncologic efficiency.

FT is based on the treatment of a part of the prostate, containing the index lesion. The index lesion is identified as a single visible lesion up to 12 mm at multiparametric MRI (mpMRI), which is biopsied with a fusion biopsy obtaining a Gleason score inferior or equal to 3+4. These features allow a focal treatment aimed to ablate the area containing the tumor. In case of a concomitant presence of 1 or 2 cores of Gleason score 3+3 found at systematic biopsy and invisible to mpMRI, a strategy of surveillance will be adopted, focusing the treatment only on the index lesion (only in patients older than 70 years old). Different sources of energy have been used to date for focal therapy. Among these, has emerged a very low loss (VLL) microwave ablation system, called TATO3®, specifically developed to work with the fusion biopsy platform Koelis Trinity® that allows an accurate 3D reconstruction of the prostate, with the goal to offer a targeted treatment after a targeted biopsy. Aim of this experimental trial is to evaluate the efficacy of the Trinity®-guided TATO3® treatment in the ablation of the index lesion, together with the safety of the procedure and the short-term oncologic outcomes.

DETAILED DESCRIPTION:
Focal therapy (FT) for prostate cancer (PCa) is an interesting therapeutic option for localized disease with a favorable low- to intermediate-risk profile. The aim of this approach is to offer a personalized and less aggressive treatment as compared to radical treatments such as radical prostatectomy (RP) or primary radiation therapy, reducing functional morbidity while maintaining oncologic efficiency.

FT is based on the treatment of a part of the prostate, containing the index lesion. Over 90% of PCa are multifocal, and unilateral disease is estimated to be present in only 20-40% of patients. Despite the multifocal nature of PCa, many affected men have just a single substantial lesion, which is called index lesion. Ohori et al determined that up to 80% of PCa volume arises through the index lesion. Clinically, vast evidence indicates that the index lesion features predict the behavior of the disease. Indeed, risk stratification of the index lesion predicts PCa outcomes, irrespectively from the presence of unilateral or bilateral disease, and most metastatic PCa arise from the cell clone of the index lesion. FT relies on the concept that residual PCa in the untreated area does not compromise long-term disease control, given that it falls into the criteria of active surveillance. The success of focal therapy strongly depends on the ability to detect the foci of PCa through multiparametric magnetic resonance imaging (mpMRI), which has gained a paramount role in PCa diagnosis. Clinically significant prostatic lesions have features detectable at mpMRI and can be targeted with fusion biopsies, which combine the data coming from mpMRI and transrectal ultrasound (TRUS) imaging. Data from PROMIS trial demonstrated MRI sensitivity of 93% for clinically significant cancer, and a meta-analysis by Moldovan et al showed a negative predictive value of mpMRI of 88.1%. A European consensus meeting suggested that mpMRI in combination of a systematic sampling achieves a negative predictive value of 90-95%. Bearing in mind the limitations of the mpMRI, however, to-date systematic biopsies are mandatory, to ensure the most accurate sampling possible, and any FT performed should consider a reasonable security margin.

For a successful treatment, patient selection is essential. Currently, the ideal candidates for FT should be patients harboring intermediate-risk PCa with favorable features and a limited component of Gleason score pattern 4. A 2015 consensus meeting stated that providing FT to patients with low-risk prostate cancer would represent overtreatment in men suitable for active surveillance. Furthermore, candidates for FT must have a life expectancy of more than 5 years and a WHO performance status of 0 or 1. In the last years, FT has solidly evolved from low-risk to intermediate-risk disease: since the first FT trials, more than 2700 patients have been treated, and this approach is now at the level of exploration of indications, quality control measures, and reproducibility in larger trials. In 2017, a randomized controlled trial (RCT) has shown the potential benefits of FT versus active surveillance in low-risk PCa in terms of cancer progression, secondary treatments, and negative biopsies at 2-yrs follow-up. In intermediate-risk PCa, another RCT of partial prostate ablation versus RP has completed the feasibility phase: the main study is set up, with the goal to prove the benefit of FT versus RP in terms of PCa mortality. In line with the recommendations of the 2015 consensus meeting, the investigators believe that suitable candidates for FT are those with a single small focus of Gleason score 7 (3+4) PCa, with possible limited adjunctive presence of clinically insignificant foci of Gleason score 6 (3+3) invisible to mpMRI. When speaking of FT for PCa, several energy modalities have been developed, including high-frequency ultrasound (HIFU), cryotherapy, laser interstitial thermotherapy, photodynamic therapy, irreversible electroporation, brachytherapy, and radiofrequency ablation. To date, studies were able to prove the feasibility, low morbidity profile, and satisfying short- and medium-term oncologic results of FT, mainly based on imaging and rebiopsy. Nevertheless, according to the last European Association of Urology (EAU) guidelines, FT is still considered experimental, to be offered within a clinical trial. Recently, among energy modalities has emerged also a very low loss (VLL) microwave ablation system, called TATO3®, specifically developed to work with the fusion biopsy platform Koelis Trinity® that allows an accurate 3D reconstruction of the prostate, with the goal to offer a targeted treatment after a targeted biopsy. Aim of this experimental trial is to evaluate the efficacy of the Trinity®-guided TATO3® treatment in the ablation of the index lesion, together with the safety of the procedure and the short-term oncologic outcomes.

Since the 1980s, microwaves have been widely used for the treatment of Benign Prostatic Hyperplasia (BPH). Low intensity energy is applied to the entire organ to reduce the volume of the gland. Several studies have shown the safety of microwaves propagation through the prostate with transurethral, transperineal and transrectal accesses, while variable results have been achieved in terms of prostate volume reduction.

The treatment of PCa by microwaves requires the use of higher energy as compared to BPH treatment, in order to irreversibly denature tumor cells. A phase I/II clinical has been led since 1998 to investigate the safety and efficacy of transperineal microwave therapy for recurrent PCa following external beam radiation therapy. A preliminary result on 25 patients has shown a very low complication rate following the treatment, and good oncological results. Six months after the treatment, 64% of the biopsy result were negative. On the last update of 2004 with 41 patients enrolled, no serious complications were observed as a result of the procedure and, although mild continence problems were encountered, these were generally temporary.

TATO3® VLL microwave ablation system represents the last evolution in the field of microwave treatment for PCa. Following dry lab testing, it has been experimented in the animal setting on dogs. More recently, it has been used at Hôpital Cochin, Paris in the setting of clinical study, where preliminary results on 10 patients with low risk PCa showed an excellent safety profile of targeted focal microwave treatment for the ablation of index tumor. Final results are awaited this summer. Another study is ongoing in at Erasme Hospital, Brussels, treating patients already scheduled for radical prostatectomy, with the aim of examining the extension of the treated area and confirming the absence of cancerous cells. To-date, the treatment is well tolerated and efficacious.

Since 2015, the investigators have acquired a significant expertise in the field of prostate fusion biopsies, achieving outstanding cancer detection rates and improving the risk stratification of newly diagnosed PCa. This expertise has been gained using different platforms in commerce, from the Koelis Urostation® to the most recent Koelis Trinity®, and the investigators have reported the outcomes of these fusion biopsies on a multicentric series of more than 2.000 patients, the largest series of fusion biopsies ever published in the literature. The natural step forward would be the implementation of the Koelis bioptic platform with the possibility of delivering a focal treatment to the foci of PCa, which can be achieved with TATO3® microwave ablation system, minimizing side effects while maintaining cancer control.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 to 80 years old, with 10 years life expectancy
* WHO Performance status 0 or 1
* Newly diagnosis of low to intermediate-risk PCa, defined by T1c or T2a clinical stage, PSA rate <20 ng/ml, unique clinically significant cancer focus visible on mpMRI, scored as ISUP grade group 1 (Gleason score 3+3) or 2 (Gleason score ≤3+4), up to 12 mm in diameter (index lesion). This focal treatment does not intend to replace active surveillance: in the cases where the indications are common to both options, focal treatment will be offered as a viable alternative to those patients unwilling to undergo active surveillance.
* All patients must have been diagnosed with transrectal or transperineal targeted and systematic biopsies performed with Koelis Trinity® system
* The presence of up to 2 additional cores of Gleason score 3+3 detected on systematic biopsies and invisible to mpMRI (therefore considered as non-significant lesions) is allowed in patients ≥70 years old: these lesions will be put under surveillance, as per regional protocol called START.
* Patient accepting to be followed after the study
* Free, informed and written consent

Exclusion Criteria:

* Past medical history of prostate radiotherapy or pelvic trauma
* Presence of other concomitant cancers
* Diagnosis of chronic prostatitis as defined by EAU guidelines
* Severe benign prostatic hyperplasia (BPH)-related lower urinary tract symptoms, defined by an IPSS score >18
* Inability to perform mpMRI
* Suspicion of extracapsular extension or seminal vesicles invasion on mpMRI
* Tumor largest axis >12 mm on mpMRI
* Distance between cancer focus and apex <5 mm on the prostate MRI
* Distance between cancer focus and rectum <5 mm on the prostate MRI
* Presence of one or more other clinically significant cancer foci, beyond the index lesion, scored as Gleason ≥7.
* Presence of more than two additional cores of Gleason score 6 (3+3) on systematic biopsies, beyond the index lesion
* Patients undergone biopsy with a system other than Koelis Trinity®
* Patients already participating in a clinical trial

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Complete tumor ablation | 6 months after treatment
  absence of tumor at the site of treatment in the repeated targeted biopsies at 6 months.

SECONDARY OUTCOMES:
Gleason score pattern 4 tumor ablation | 6 months after treatment
  absence of tumor Gleason score pattern 4 at the site of treatment in the repeated targeted biopsies at 6 months
Functional score IPSS | 1 week, 1 month, 3 months, 6 months after treatment
  change in the functional score IPSS (International Prostate Symptom Score, from 0 (best) to 35 (worse)) 1 week, 1 month, 3 months and 6 months after the treatment, as compared to the basal score before focal therapy
Functional score IIEF-5 | 1 week, 1 month, 3 months, 6 months after treatment
  change in the functional score IIEF-5 (International International Index of Erectile Function-5 score, from 5 (worse) to 25 (best)) 1 week, 1 month, 3 months and 6 months after the treatment, as compared to the basal score before focal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marco Oderda, MD, PhD, Principal Investigator — A.O.U. Città della Salute e della Scienza di Torino
Locations (1):
- A.O.U. San Giovanni Battista Molinette, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanchez-Salas R, de la Rosette J, Polascik TJ, Carneiro A, Sivaraman A, Cathelineau X, Walz J. Focal Therapy for Prostate Cancer: A More Vehement View of the Approach Could Translate into Real Benefits for Our Patients. Eur Urol. 2018 Nov;74(5):537-539. doi: 10.1016/j.eururo.2018.04.018. Epub 2018 May 1. PMID 29724502
- [Result] Barbalias GA, Liatsikos EN. Transrectal microwave hyperthermia for patients with benign prostatic hyperplasia. Int J Urol. 1998 Mar;5(2):157-62. doi: 10.1111/j.1442-2042.1998.tb00267.x. PMID 9559842
- [Result] Sherar MD, Gertner MR, Yue CK, O'Malley ME, Toi A, Gladman AS, Davidson SR, Trachtenberg J. Interstitial microwave thermal therapy for prostate cancer: method of treatment and results of a phase I/II trial. J Urol. 2001 Nov;166(5):1707-14. doi: 10.1016/s0022-5347(05)65658-3. PMID 11586207
- [Result] Oderda M, Marra G, Albisinni S, Altobelli E, Baco E, Beatrici V, Cantiani A, Carbone A, Ciccariello M, Descotes JL, Dubreuil-Chambardel M, Eldred-Evans D, Fasolis G, Ferriero M, Fiard G, Forte V, Giacobbe A, Kumar P, Lacetera V, Mozer P, Muto G, Papalia R, Pastore A, Peltier A, Piechaud T, Simone G, Roche JB, Roupret M, Rouviere O, Van Velthoven R, Gontero P. Accuracy of elastic fusion biopsy in daily practice: Results of a multicenter study of 2115 patients. Int J Urol. 2018 Dec;25(12):990-997. doi: 10.1111/iju.13796. Epub 2018 Sep 5. PMID 30187529
- [Result] Schepps JL, Foster KR. The UHF and microwave dielectric properties of normal and tumour tissues: variation in dielectric properties with tissue water content. Phys Med Biol. 1980 Nov;25(6):1149-59. doi: 10.1088/0031-9155/25/6/012. PMID 7208627